CLINICAL TRIAL: NCT01981330
Title: Pilot Study of Patients With Severe Hoarseness and Vocal Fold Scarring Treated With Mesenchymal Stem Cells With and Without Hyaluronan Gel
Brief Title: Pilot Study of Stem Cell Treatment of Patients With Vocal Fold Scarring
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: The Swedish Research Council (Other Government); Laryngfonden (Unknown); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Stellan Hertegård, MD PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/1650 and 2014-51432
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Improved Healing of Scarred Vocal Folds; Improved Vocal Fold Status; Improved Vocal Fold Function
Keywords: vocal fold scarring; mesenchymal stem cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aMSC with and without hyaluronan gel (Experimental): autologous mesenchymal stem cells (aMSC) injected into the vocal folds in 8 patients and aMSC mixed with hyaluronan gel in 8 patients
  Interventions: Biological: aMSC; Biological: aMSC+hyaluronan gel

INTERVENTIONS:
Biological: aMSC — aMSC injected into the vocal fold of the patient
Biological: aMSC+hyaluronan gel — aMSC+ hyaluronan gel is injected into the patients vocal fold

SUMMARY:
This is a pilot-study of 16 selected Swedish patients which all have severe hoarseness or aphonia due to vocal fold scarring (from previous surgery, radiation therapy, inflammation or possibly hereditary). The patients are operated with phonomicrosurgical dissection of the scarred vocal folds, removal or scar tissue and injection of autologous mesenchymal stroma cells, aMSC (which were previously harvested from each patients´s bone marrow, purified, expanded and characterized according to standard procedure at the Center of Hematology and Regenerative Medicine Karolinska University Hospital Huddinge). 8 Patients is planned to be treated with a single injection of aMSC and 8 patients with injection of aMSC mixed with a carrier hyaluronan gel developed at Uppsala University Sweden and at the Karolinska Institute. The laryngeal status, vocal fold function, and voice function will be followed individually with an advanced battery of examinations performed before and up to 1 year postoperatively. Side effects and complications are noted and reported during surgery and following surgery at regular intervals during at least 1 year Since spring 2015 no new patients have been recruited and no treatments are given during 2016 or 2017. The monitoring authority was changed from Swedish National Board of Health to Swedish Medical Product Agency (MPA) in March/April 2016. Further inclusions and treatments are postponed until permission is granted from MPA to continue the study.

ELIGIBILITY:
Inclusion Criteria:

* severe hoarseness
* vocal fold scarring
* no active other treatment
* age above 18 years

Exclusion Criteria:

* active treatment of laryngeal disorder
* active inflammatory condition of the larynx
* diagnosed or suspicions of local malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Improved healing of scarred vocal folds | 1 year postoperatively
  Laryngeal and general ear, nose, and throat status will be followed for each patient at least one year after primary treatment. This includes examination of signs of local (laryngeal) inflammatory reaction/defect healing, e.g. polyp or granuloma formation, inflammatory reaction after local aMSC injection It also includes repetitive examinations of vocal fold function and voice function including high speed examination of the vocal folds, acoustic voice analysis and phonation pressure measurements as well as subjective ratings by means of Voice handicap index scale

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Hertegard S, Nagubothu SR, Malmstrom E, LeBlanc K. Treatment of vocal fold scarring with autologous bone marrow-derived human mesenchymal stromal cells-first phase I/II human clinical study. Stem Cell Res Ther. 2020 Mar 20;11(1):128. doi: 10.1186/s13287-020-01632-8. PMID 32197630